CLINICAL TRIAL: NCT00193947
Title: An Evaluation of the Development of Nevirapine Induced Mutations in HIV Patients Initiating or Discontinuing Combination Antiretroviral Therapy
Status: Terminated | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: University Health Network Toronto, university health network
Other Study IDs: 03-0162-B
Record Dates: First submitted 2005-09-15; First posted 2005-09-19 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2007-04

CONDITIONS: Drug Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- women initiating ARV therapy during pregnancy with neveripine

SUMMARY:
Hypothesis

Nevirapine resistance developed in women and infants in the HIVNET 006 and 012 cohorts as a consequence of use of an agent with a long t½ as monotherapy in individuals with high viral loads.

Objective 1 To demonstrate that Nevirapine resistance does not develop in HIV infected patients when used as part of triple antiretroviral combination therapy between the initiation of treatment and suppression of HIV RNA to <1000 copies/ml.

Objective 2 To demonstrate that resistance to nevirapine does not develop when patients with suppressed HIV RNA discontinue combination antiretroviral therapy which contains nevirapine.

DETAILED DESCRIPTION:
The HIVNET 012 clinical trial demonstrates a cost effective strategy to prevent maternal fetal transmission of HIV. In this study, a single 200 mg dose of Nevirapine was given to pregnant Ugandan women at the onset of labour and a single 2 mg/kg dose to their infants within 72 hours of birth (1). Given the efficacy, simplicity and low cost of this regime, the World Health Organization recently recommended implementation of this regimen as one of several options for prevention of maternal fetal transmission of HIV in resource limited settings.

Pharmacokinetic studies have demonstrated that 200 mg of Nevirapine given to the mother during labour results in concentrations >100 mg/mL (10 times the in vitro IC50) in the newborn. Nevirapine elimination is prolonged in both mothers and infants with median t½ of 36.8 to 65.7 hours. Administration of 200 mg orally to the mother and a single 2 mg/kg oral dose to the infant at 48-72 hours, maintains serum concentration in the infants >100 mg/ml through 7 days of life (2, 3)

Early studies demonstrated that the use of Nevirapine monotherapy resulted in a rapid selection of Nevirapine resistant mutations (4). This was associated with loss of antiviral activity and return of the viral load to baseline within 12 weeks. It appeared very soon that the non-nucleoside reverse transcriptase inhibitors were drugs with a low genetic barrier and that a single mutation in the reverse transcriptase gene induced a high level of phenotypic resistance (5). Similarly, when Nevirapine was used in combination with a single nucleoside, and there was incomplete suppression of viral replication, resistance emerged to the non-nucleoside reverse transcriptase inhibitor (6).

In contrast, when used as part of triple antiretroviral combination and there was successful inhibition of viral replication to <50 copies/ml, the viral response was maintained in 50% of patients out to 48 weeks (7, 8, 9, 10). However, again when virologic control is lost, resistance to Nevirapine emerges rapidly in 50-100% of patients (11). It is unclear whether or not these mutations developed during the initial suppression of viral load replication or during rebound of viremia with failure.

Given the pharmacokinetics of Nevirapine in pregnant women and infants, concern was raised that mother and child would be exposed to Nevirapine monotherapy for one to several days and that the selection of resistant mutants could arise limiting this strategy over the long term. In fact, a recent sub-analysis of the HIVNET 012 cohort found Nevirapine resistant mutations in 21/111 (19%) of women tested at 6-8 weeks after delivery. The K103N was the most common mutation. Women with the highest baseline viral load developed the mutations more frequently. Nevirapine resistant mutations were also detected in 11/24 or (46%) of infected infants at 6-8 weeks. In contrast to the mothers, the Y181C was the most commonly detected.

Similarly, the K103N resistance mutation was detected 6 weeks after Nevirapine administration in 3/15 (20%) women in the HIVNET006 phase I/II trial. This had the same Nevirapine dosing schedule as HIVNET012 (12).

New information has become available based on recent post-marketing surveillance data clarifying risk factors for severe life threatening and fatal hepatotoxicity with nevirapine. Women with CD4 counts > 250 cellsmm3 at initiation of therapy including pregnant women receiving chronic treatment for HIV infection are at considerably higher risk (12-fold) of hepatotoxicity which in some cases has been fatal. The greatest risk of severe and potentially fatal hepatic events occurs in the first 6 weeks of therapy. However, the risk continues after this time and patients should be closely monitored for the first 18 weeks of therapy. For this reason, women with CD4 > 250/mm3 will not be included in Objective 1 of this study.

Hypothesis

Nevirapine resistance developed in women and infants in the HIVNET 006 and 012 cohorts as a consequence of use of an agent with a long t½ as monotherapy in individuals with high viral loads.

Objective 1 To demonstrate that Nevirapine resistance does not develop in HIV infected patients when used as part of triple antiretroviral combination therapy between the initiation of treatment and suppression of HIV RNA to <1000 copies/ml.

Objective 2 To demonstrate that resistance to nevirapine does not develop when patients with suppressed HIV RNA discontinue combination antiretroviral therapy which contains nevirapine.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria (Objective 1)

1. HIV infected adults
2. Antiretroviral naïve
3. Viral load >1000 copies/ml
4. Initiating combination antiretroviral therapy, which includes nevirapine.

Exclusion Criteria (Objective 1)

1. Women with CD4 counts > 250/mm3

Inclusion Criteria (Objective 2)

1. HIV infected adults
2. On their initial ARV combination which contains nevirapine
3. HIV RNA < 50 copies/ml
4. Decision to discontinue ARV therapy at the completion of pregnancy or for a drug holiday
5. Not resistant to nevirapine.

Note that since most patients meeting the criteria for Objective 1 are expected to achieve HIV RNA < 50 copies/mL, the patient populations for Objectives 1 and 2 will be almost the same.

-

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women attending the UHN immunodeficiency clinic
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2003-11; Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To demonstrate that Nevirapine resistance does not develop in HIV infected patients when used as part of triple antiretroviral combination therapy between the initiation of treatment and suppression of HIV RNA to <1000 copies/ml. | during viral suppression

SECONDARY OUTCOMES:
to determine whether ARV resistance emerges when pregnant women discontinue ARV | 6 months after drug discontinutation or until viral rebound

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Walsmley, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada